CLINICAL TRIAL: NCT04822922
Title: Safety of Human Umbilical Cord-derived Mesenchymal Stem Cell (UC-MSC) Transfusion for Acute-on-chronic Liver Failure Patients
Brief Title: Safety of UC-MSC Transfusion for ACLF Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hai Li (Other)
Responsible Party: Sponsor-Investigator, Hai Li, chief physician of gastroenterological division, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-ACLF-1
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: ACLF; mesenchymal stem cell; safety
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Intervention Model Description: 3 parallel group with different doses of UC-MSC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose (Experimental): hUC-MSCs 4*10^5/kg/each time
  Interventions: Genetic: Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs)
- middle dose (Experimental): hUC-MSCs 8*10^5/kg/each time
  Interventions: Genetic: Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs)
- high dose (Experimental): hUC-MSCs 12*10^5/kg/each time
  Interventions: Genetic: Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs)

INTERVENTIONS:
Genetic: Human umbilical cord-derived mesenchymal stem cells (hUC-MSCs) — The hUC-MSCs were injected intravenously on the 1, 4, 7 and 10 days after patients recruitment. The treatment doses include low dose: 4*10^5 cells/kg/each time, and medium dose: 8*10^5 cells/kg/each time, high dose 12*10^5 cells/kg/each time. After 3 groups of patients were enrolled, the group with appropriate safety and effectiveness was selected and the other 4 subjects were included.

SUMMARY:
Acute on chronic liver failure (ACLF) is a type of critically ill liver disease with high short-term mortality in liver disease. Liver transplantation is currently the only method to improve survival. Current clinical research evidence shows that mesenchymal stem cells can reduce the mortality of ACLF patients and are safe. This study aims to explore the safety of umbilical cord mesenchymal stem cells (UC-MSCs) in the treatment of ACLF. The study population is ACLF patients with 1-2 organ failures. To explore the safety of 3 doses of UC-MSCs, 16 patients need to be enrolled. The main observation indicators are the short-term and long-term safety of the treatment. All patients need to receive the standard medical treatment (SMT) at the same time. Stem cell treatment is given by intravenous infusion on the first, fourth, seventh, and tenth day. The occurrence of adverse events (AE) and serious adverse events(SAE) before and after the infusion will be observed. After the patient is discharged from the hospital, patients will be followed , the follow-up time is 5 years.

DETAILED DESCRIPTION:
Acute-on-chronic liver failure (acute-on-chronic liver failure, ACLF) is a special type of rapid deterioration of liver function that occurs on the basis of cirrhosis or non-cirrhosis, which is characterized by sequential multiple organ failure and high short-term (28 days) mortality (15%). ACLF was first proposed by Jalan R and Williams R. in 2002. It is a newly discovered type of critically ill liver disease characterized by high short-term mortality after hospitalization [1]. At present, the pathophysiological mechanism of ACLF is not clear, and its definition in Europe and Asia-Pacific is still controversial. However, severe systemic inflammatory response is often closely related to the cause, accompanied by single or multiple organ failure are three important characteristics of ACLF. In the past ten years, the prevalence of ACLF has increased. Due to the rapid progress of the disease and the close relationship between mortality and organ failure, there is no effective method to improve the survival rate of ACLF patients except liver transplantation. The latest literature review shows that the 28-day and 90-day mortality rates are as high as 27.8-37.6% and 40-, respectively. 51.2%[2].

In 2013, European Association for the Study of Chronic Acute Liver Failure（EASL-CLIF） conducted a prospective multi-center EASL-CLIF Chronic Acute Liver Failure (CANONIC) study in 29 liver disease treatment centers in eight European countries, and proposed chronic liver failure-sequential organ failure assessment（CLIF-SOFA）score is used as the clinical diagnostic criteria for alcoholic and hepatitis B virus（HBV）related ACLF. According to the CLIF-SOFA score, the 90-day mortality rate of ACLF patients is as high as 51%, while that of non-ACLF patients is 10% [3]. The European CANONIC study also shows that systemic inflammation is the main driving force of multiple organ failure, which is a typical pathogenesis of ACLF patients with western liver cirrhosis [4]. For another, the current Asian ACLF diagnostic criteria is the Asia Pacific Association for the Study of Liver Diseases (APASL) criteria, which reached a consensus in 2009, and the guidelines were improved in 2014, but there is still a lack of multi-center, prospective evidence-based medical evidence to support . In 2016, led by the person in charge of this project, an oriental ACLF prospective multi-center observation cohort was established in China, which included 3970 ACLF high-risk patients, filling the gap in the natural course and mortality of oriental ACLF patients, and established a 90-day oriental ACLF diagnostic criteria for mortality [5]. The person in charge of this project also explored the pathophysiological mechanism of ACLF patients in areas with high prevalence of oriental HBV. The study showed that submassive hepatic necrosis is an important histological feature in ACLF patients with HBV-related cirrhosis. The systemic inflammatory response of multiple organ failure caused by parenchymal liver cells has a similar mechanism to that of western alcoholic ACLF [6]. Although the causes of ACLF type are not the same in the East and the West, the cohorts from the East and the West have confirmed the short-term high mortality rate of ACLF. Systemic inflammation, sub-large necrosis, and aseptic inflammation may all important reasons that lead to multiple organ failure and eventual death of ACLF patients.

Due to the high short-term mortality of ACLF and the limited liver source for liver transplantation, exploring new methods for the treatment of ACLF is a major issue facing clinical research. Mesenchymal stem cells have great application prospects in regenerative medicine because of their strong self-renewal, low immunogenicity, non-tumorigenicity and strong immune regulation ability[7]. Many previous documents have confirmed that mesenchymal stem cells in animal models can promote liver cell regeneration, resist inflammation, regulate local microenvironment and anti-fibrosis [8-10]. Among them, umbilical cord mesenchymal stem cells (UC-MSC) have attracted attention of researchers because they are easily obtained from the medical waste-the umbilical cord, are not invasive, and have high expansion capabilities in vitro [11]. The possible mechanism of UC-MSC in the treatment of end-stage liver disease is that it can repair the liver. At present, there are the following opinions: ① Cell rehabilitation. In the case of liver failure, MSC can differentiate into hepatocytes and play an alternative therapeutic effect. A large number of studies have shown that MSC can be differentiated into functional hepatocytes in different inducing factors and culture systems in vitro, capable of storing glycogen and urea synthesis. Function; ②Immune regulation. Studies have shown that MSC can regulate immune cells by secreting a variety of cytokines in the body, and play an immunomodulatory effect; ③Anti-fibrosis. MSC can induce hepatic stellate cell apoptosis or inhibit its activation, and can secrete anti-fibrotic substances such as granulocyte colony stimulating factor and matrix metallopeptidase 9（MMP-9）to reduce the deposition of extracellular matrix and inhibit the formation of liver fibrosis.

According to the results of a single-center clinical trial published by the Third Affiliated Hospital of Sun Yat-sen University in the previous period, there were no serious adverse reactions at 6 hours and 72 weeks after intravenous infusion of MSCs. The dose was (1-6)*10^7 cells/time for 4 times, confirming the safety and effectiveness of both low-dose and high-dose treatments. Another open clinical trial of Beijing 302 Hospital used mesenchymal stem cells at a dose of 5*10^5 cells/kg (based on the patient's weight of 60kg, the dose was 3*10^7 cells/time), excluded severe ACLF patients accompanied by severe infections and other sever complications. In addition, previous pharmacokinetic tests showed that the half-life of mesenchymal stem cells in animals is 3 days.

Therefore, this research plans to carry out a single-center open clinical trial to confirm the safety of umbilical cord-derived mesenchymal stem cells in the treatment of ACLF, and provide stronger clinical evidence for the safety of UC-MSCs in the treatment of ACLF.

ELIGIBILITY:
Inclusion Criteria:

1. . Age 18-70 years old;
2. . A history of chronic liver disease, chronic acute liver failure (ACLF) caused by various causes, 1-2 organ failure (ACLF diagnosis is based on the European EASL diagnostic criteria, and the organ failure criteria is based on CLIF-OF);
3. . The patient or adult family members agree to participate in this study and sign an informed consent form;

Exclusion Criteria:

* Those who meet any of the following conditions will not be included:

  1. Those who intend to undergo artificial liver treatment;
  2. Those who have received liver transplantation and any form of stem cell therapy;
  3. Malignant tumors in or outside the liver; or imaging findings suggest malignant mass in the liver or tuberculosis;
  4. Complicated with severe autoimmune diseases; combined with severe cardiopulmonary insufficiency; renal replacement therapy; Immunosuppressive therapy; HIV/tuberculosis infection; alcohol/drug addiction; participated in drug trials in the past 3 months;
  5. Gastrointestinal bleeding or serious infection occurred in the past one month;
  6. Pregnant and lactating women;
  7. Those who do not have the ability to make independent judgments and have no direct adult family members to sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2024-07-21 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment | 1 month since intervention start
  The purpose of this trial is to observe the short-term safety of low, medium and high doses of hUC-MSCs in the treatment of ACLF patients. The primary endpoint of the study was serious adverse events that occurred during the course of one month of treatment. If serious adverse reactions(SAE) occur during the treatment in hospital, the intervention will be stopped and the study will be terminated.

SECONDARY OUTCOMES:
Short-time efficacy of treatment | 90 days
  To assess the efficacy of hUC-MSCs in the treatment of ACLF patients, patients will be followed-up, and the prognosis at each time point will be collected as our schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Hai Li, Study Director — Digestive Department of Renji Hospital,Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao TongUniversity,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreau R, Jalan R, Gines P, Pavesi M, Angeli P, Cordoba J, Durand F, Gustot T, Saliba F, Domenicali M, Gerbes A, Wendon J, Alessandria C, Laleman W, Zeuzem S, Trebicka J, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Acute-on-chronic liver failure is a distinct syndrome that develops in patients with acute decompensation of cirrhosis. Gastroenterology. 2013 Jun;144(7):1426-37, 1437.e1-9. doi: 10.1053/j.gastro.2013.02.042. Epub 2013 Mar 6. PMID 23474284
- [Background] Arroyo V, Moreau R, Jalan R. Acute-on-Chronic Liver Failure. N Engl J Med. 2020 May 28;382(22):2137-2145. doi: 10.1056/NEJMra1914900. No abstract available. PMID 32459924
- [Background] Claria J, Stauber RE, Coenraad MJ, Moreau R, Jalan R, Pavesi M, Amoros A, Titos E, Alcaraz-Quiles J, Oettl K, Morales-Ruiz M, Angeli P, Domenicali M, Alessandria C, Gerbes A, Wendon J, Nevens F, Trebicka J, Laleman W, Saliba F, Welzel TM, Albillos A, Gustot T, Benten D, Durand F, Gines P, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium and the European Foundation for the Study of Chronic Liver Failure (EF-CLIF). Systemic inflammation in decompensated cirrhosis: Characterization and role in acute-on-chronic liver failure. Hepatology. 2016 Oct;64(4):1249-64. doi: 10.1002/hep.28740. Epub 2016 Aug 25. PMID 27483394
- [Background] Gu WY, Xu BY, Zheng X, Chen J, Wang XB, Huang Y, Gao YH, Meng ZJ, Qian ZP, Liu F, Lu XB, Shang J, Li H, Wang SY, Sun X, Li H. Acute-on-Chronic Liver Failure in China: Rationale for Developing a Patient Registry and Baseline Characteristics. Am J Epidemiol. 2018 Sep 1;187(9):1829-1839. doi: 10.1093/aje/kwy083. PMID 29762630
- [Background] Li H, Xia Q, Zeng B, Li ST, Liu H, Li Q, Li J, Yang SY, Dong XJ, Gao T, Munker S, Liu Y, Liebe R, Xue F, Li QG, Chen XS, Liu Q, Zeng H, Wang JY, Xie Q, Meng QH, Wang JF, Mertens PR, Lammert F, Singer MV, Dooley S, Ebert MP, Qiu DK, Wang TL, Weng HL. Submassive hepatic necrosis distinguishes HBV-associated acute on chronic liver failure from cirrhotic patients with acute decompensation. J Hepatol. 2015 Jul;63(1):50-9. doi: 10.1016/j.jhep.2015.01.029. Epub 2015 Jan 31. PMID 25646889
- [Background] Galipeau J, Sensebe L. Mesenchymal Stromal Cells: Clinical Challenges and Therapeutic Opportunities. Cell Stem Cell. 2018 Jun 1;22(6):824-833. doi: 10.1016/j.stem.2018.05.004. PMID 29859173
- [Background] Arthur MJ. Reversibility of liver fibrosis and cirrhosis following treatment for hepatitis C. Gastroenterology. 2002 May;122(5):1525-8. doi: 10.1053/gast.2002.33367. No abstract available. PMID 11984538
- [Background] Cho KA, Lim GW, Joo SY, Woo SY, Seoh JY, Cho SJ, Han HS, Ryu KH. Transplantation of bone marrow cells reduces CCl4 -induced liver fibrosis in mice. Liver Int. 2011 Aug;31(7):932-9. doi: 10.1111/j.1478-3231.2010.02364.x. Epub 2010 Nov 24. PMID 21092070
- [Background] Aurich I, Mueller LP, Aurich H, Luetzkendorf J, Tisljar K, Dollinger MM, Schormann W, Walldorf J, Hengstler JG, Fleig WE, Christ B. Functional integration of hepatocytes derived from human mesenchymal stem cells into mouse livers. Gut. 2007 Mar;56(3):405-15. doi: 10.1136/gut.2005.090050. Epub 2006 Aug 23. PMID 16928726
- [Background] Arutyunyan I, Elchaninov A, Makarov A, Fatkhudinov T. Umbilical Cord as Prospective Source for Mesenchymal Stem Cell-Based Therapy. Stem Cells Int. 2016;2016:6901286. doi: 10.1155/2016/6901286. Epub 2016 Aug 29. PMID 27651799
- [Background] Xue R, Meng Q, Li J, Wu J, Yao Q, Yu H, Zhu Y. The assessment of multipotent cell transplantation in acute-on-chronic liver failure: a systematic review and meta-analysis. Transl Res. 2018 Oct;200:65-80. doi: 10.1016/j.trsl.2018.05.006. Epub 2018 Jun 23. PMID 30016629
- [Background] Xue R, Meng Q, Dong J, Li J, Yao Q, Zhu Y, Yu H. Clinical performance of stem cell therapy in patients with acute-on-chronic liver failure: a systematic review and meta-analysis. J Transl Med. 2018 May 10;16(1):126. doi: 10.1186/s12967-018-1464-0. PMID 29747694
- [Background] Chen B, Wang YH, Qian JQ, Wu DB, Chen EQ, Tang H. Human mesenchymal stem cells for hepatitis B virus-related acute-on-chronic liver failure: a systematic review with meta-analysis. Eur J Gastroenterol Hepatol. 2018 Oct;30(10):1224-1229. doi: 10.1097/MEG.0000000000001156. PMID 29727380
- [Background] Peng L, Xie DY, Lin BL, Liu J, Zhu HP, Xie C, Zheng YB, Gao ZL. Autologous bone marrow mesenchymal stem cell transplantation in liver failure patients caused by hepatitis B: short-term and long-term outcomes. Hepatology. 2011 Sep 2;54(3):820-8. doi: 10.1002/hep.24434. Epub 2011 Jul 14. PMID 21608000
- [Background] Lin BL, Chen JF, Qiu WH, Wang KW, Xie DY, Chen XY, Liu QL, Peng L, Li JG, Mei YY, Weng WZ, Peng YW, Cao HJ, Xie JQ, Xie SB, Xiang AP, Gao ZL. Allogeneic bone marrow-derived mesenchymal stromal cells for hepatitis B virus-related acute-on-chronic liver failure: A randomized controlled trial. Hepatology. 2017 Jul;66(1):209-219. doi: 10.1002/hep.29189. Epub 2017 May 27. PMID 28370357
- [Background] Shi M, Zhang Z, Xu R, Lin H, Fu J, Zou Z, Zhang A, Shi J, Chen L, Lv S, He W, Geng H, Jin L, Liu Z, Wang FS. Human mesenchymal stem cell transfusion is safe and improves liver function in acute-on-chronic liver failure patients. Stem Cells Transl Med. 2012 Oct;1(10):725-31. doi: 10.5966/sctm.2012-0034. Epub 2012 Oct 11. PMID 23197664